CLINICAL TRIAL: NCT05239507
Title: A Multicountry, Multicentre, Noninterventional, Retrospective Study to Describe the Real-world Management Outcomes in Patients With Unresectable Hepatocellular Carcinoma
Brief Title: OREIOS International Study
Acronym: OREIOS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D419CR00025
Record Dates: First submitted 2021-11-30; First posted 2022-02-15 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Considering the treatment landscape with its dynamic algorithms and new approaches of sequencing, it is important to identify patient management patterns and survival outcomes arising from the current standard of care. Based on all these considerations, this multicountry, multicentre, noninterventional, real-world, retrospective study is designed to describe the management patterns, clinical characteristics, possible predictors, and survival outcomes in patients with unresectable HCC. The results of this study might help oncologists in optimal patient selection and sequencing of the systemic therapies.

DETAILED DESCRIPTION:
Patients with unresectable HCC are an extremely heterogeneous population, with several coexisting risk factors like underlying hepatic dysfunction, extrahepatic metastases, and macrovascular invasion (MVI) posing a challenge for optimum sequencing of the existing, newly approved, and emerging targeted therapies. Real-world studies have identified factors such as performance status, Child-Pugh class, MVI or extrahepatic metastasis and AFP levels, which predict the response to treatment. More than half of patients with HCC present with intermediate or advanced-stage disease (BCLC stage B, C or D) and require palliative care. Very few studies have identified the predictors of survival in advanced HCC and further exploration is warranted to optimize treatment regimen. Systemic therapy based on multi-kinase inhibitors, anti-angiogenesis agents, and immunotherapy have become the cornerstone of advanced HCC management. Despite these advances, patients with HCC still have a poor long-term prognosis of -12 month. Clinical decision making has become challenging in cases with localized but unresectable disease or in the presence of impaired liver function; there are multiple treatment options and selection between them is not supported by direct comparative evidence. Furthermore, disease and patient characteristics seen in clinical practice may be very different from those included in clinical trials; there may be less rigorous follow up and patient counselling resulting in reduced compliance with treatments. Considering the treatment landscape with its dynamic algorithms and new approaches of sequencing, it is important to identify patient management patterns and survival outcomes arising from the current standard of care. Based on all these considerations, this multi-country, multicenter, noninterventional, real-world, retrospective study is designed to describe the management patterns, clinical characteristics, possible predictors, and survival outcomes in patients with unresectable HCC. The results of this study might help oncologists in optimal patient selection and sequencing of the systemic therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Adult female or male patients aged ≥18 years or 'adults' according to the age of majority as defined by the local regulations at index diagnosis
2. Patients or legal representative (unless a waiver is granted) willing and be able to provide informed consent according to local regulations. For deceased patients at study entry, informed consent is not mandatory.
3. Patients with radiologically or histopathologically confirmed diagnosis (at index date) of unresectable BCLC stage B HCC, not considered eligible for initial loco-regional therapya or stage C advanced or metastatic disease, between 01 January 2017 and 31 December 2019.
4. Availability of at least 12 months of follow-up data (from the index date) in the medical records at the participating site, unless patient died within the first 12 months of diagnosis.

Exclusion Criteria:

1. Patients with BCLC stage D HCC at index diagnosis
2. Patients with concomitant cancer, at the time of diagnosis of unresectable HCC, except for the nonmetastatic nonmelanoma skin cancers or in situ or benign neoplasms; a cancer is considered concomitant if it occurs within 5 years of HCC diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include patients diagnosed with unresectable HCC, who have been treated or are currently receiving treatment outside North America and Europe. Participating countries will include Brazil, Hong Kong, Oman, Kuwait, Qatar, South Korea, Russia, UAE, Saudi Arabia, Egypt, India, and Taiwan.
Sampling Method: Non-Probability Sample
Enrollment: 1127 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-03-12 (Actual); Study Completion 2023-03-12 (Actual)

PRIMARY OUTCOMES:
To describe the OS rate in patients with unresectable HCC including estimates of survival rates at 6, 12, and 18 months and at 2 years | Change from Baseline in Survival Rates at 2 years
  OS Kaplan-Meier (KM) curve and survival rates at 6, 12, and 18 months and at 2 years

SECONDARY OUTCOMES:
To describe the management patterns in patients with unresectable HCC | through study completion, an average of 2 year
  Percentage of patients receiving standard regimens alone or in combination with other systemic agents in each line of therapy (LOT)
To describe the demographic and clinical characteristics of patients with unresectable HCC | At baseline
  Demographic and clinical characteristics of patients with unresectable HCC

OTHER OUTCOMES:
To describe the survival outcomes associated with different treatment regimens for unresectable HCC | through study completion, an average of 2 year
  Survival outcomes associated with different treatment regimens for unresectable HCC
To estimate the effectiveness of different treatment regimens for unresectable HCC including real-world objective response rate (rwORR) | through study completion, an average of 2 year
  Effectiveness of different treatment regimens for unresectable HCC
To estimate the effectiveness of different treatment regimens for unresectable HCC including real-world disease control rate (rwDCR) | through study completion, an average of 2 year
  Effectiveness of different treatment regimens for unresectable HCC
To investigate the correlation between survival outcomes and clinical characteristics, liver function, and underlying disease in unresectable HCC | through study completion, an average of 2 year
  Identification of potential factors correlating with OS (median OS) among the following clinico-pathological variables:

CONTACTS AND LOCATIONS:
Locations (21):
- Brazil (2):
  - Research Site, Porto Alegre, Rio Grande do Sul
  - Research Site, São Paulo
- Egypt (4):
  - Research Site, Alexandira
  - Research Site, Asyut
  - Research Site, Cairo
  - Research Site, Menufia
- Research Site, Hong Kong, Hong Kong
- India (4):
  - Research Site, Faridabad
  - Research Site, Howrah
  - Research Site, Kolkata
  - Research Site, New Delhi
- Research Site, Kuwait City, Kuwait
- Research Site, Muscat, Oman
- Russia (3):
  - Research Site, Chelyabinsk
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- Saudi Arabia (2):
  - Research Site, Mecca
  - Research Site, Riyadh
- Research Site, Singapore, Singapore
- Research Site, Seoul, South Korea
- Research Site, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: CSR_Synopsis_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D419CR00025&attachmentIdentifier=f1902138-7446-4a1d-96fc-116805969d9c&fileName=CSR_Synopsis_Redacted.pdf&versionIdentifier=